CLINICAL TRIAL: NCT06580756
Title: Development and Validation of a Short Training Course to Help Primary Care Healthcare Professionals Identify Addictive Disorders
Brief Title: Problematic Use and Addiction in Primary Care
Acronym: PAPRICA
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: DR230127-PAPRICA
Record Dates: First submitted 2024-08-22; First posted 2024-08-30 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Addiction Disorders; Primary Care
Keywords: short training program

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group intervention: Group with a brief training
  Interventions: Other: Short training program
- group control: Group without a brief training

INTERVENTIONS:
Other: Short training program — Training in the early identification of addictive disorders in primary care
  Groups: group intervention

SUMMARY:
The morbi-mortality and social cost of addictive disorders led the French authorities to set up a government plan in 2018 to combat drugs and addictive behavior (Interministerial mission to combat drugs and addictive behaviour - (MILDECA)). In particular, it encourages early detection, which is the first stage in a validated global approach to the management of addictive disorders. Improving early identification of addictive disorders in primary care would reduce morbidity and mortality and improve quality of life for patients with addictive disorders. The identification of use disorders should be systematic in primary care and was the subject of a recommendation in 2015. Numerous tests are cited in these recommendations, but few have actually been validated in primary care, and none has been shown to be feasible. For example, only 23% of GPs claim to systematically identify alcohol consumption.

Other primary care professionals (physiotherapists, nurses, midwives, dentists, pharmacists) also have a role to play in identifying addictive disorders. The evolution of their respective professions (delegation of tasks, creation of the profession of advanced practice nurse, medical assistants) and the recent reorganization of the practice framework, both in terms of practice structures and professional community organizations, involve them in a global multidisciplinary collaboration on patient care, particularly in the early identification of addictive disorders.

The hypothesis is that the difficulties in implementing tests to identify addictive disorders in primary care are linked to the lack of specific consideration of the needs of primary care patients and caregivers.

The overall aim of the study is to improve the early detection of addictive disorders through brief training for primary care healthcare professionals.

DETAILED DESCRIPTION:
The project comprises three successive stages:

1. Design a training program with content tailored to primary care professionals;
2. Evaluate the feasibility and acceptability of the training;
3. Evaluate the implementation of this training program by comparing the incidence of addiction disorder detection by primary care professionals between a trained and an untrained group.

ELIGIBILITY:
Inclusion Criteria:

* be a primary care professional (physiotherapists, nurses, midwives, dentists, pharmacists, General practitioner)
* in ambulatory practice. Recruitment will be carried out with the help of territorial professional health communities, to include practitioners practicing in conditions representative of the diversity of primary care practice.

GPs agreeing to take part will be divided into a control group and an intervention group, by drawing lots.

Exclusion Criteria:

* Refusal to participate.
* The same participant may not be included in more than one stage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care ambulatory professional
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Number of patients who received information about the addictive disorders from the primary care professional | 24 months
  The main aim of the study was to measure the effect of brief training in the identification of addictive disorders on the rate of patients who actually received the information from the primary care professional.
number of patients identified with an addictive disorder from the primary care professional | 24 months
  The main aim of the study was to measure the effect of brief training in the identification of addictive disorders on the rate of patients who actually received the information from the primary care professional.

SECONDARY OUTCOMES:
prevalence of addictive disorders in primary care | 24 months
  Measure the prevalence
types of addictive disorders | 24 months
  List of addictive disorders identified in patients

CONTACTS AND LOCATIONS:
Overall Officials: Maxime PAUTRAT, Principal Investigator — Tours university
Locations (3):
- France (3):
  - CPTS Lanmeur, Lanmeur
  - CPTS Sud Lochois, Ligueil
  - CPTS du Vendomois, Vendôme

IPD SHARING:
Plan to Share IPD: Undecided